CLINICAL TRIAL: NCT02331394
Title: A Feasibility Study of Chinese Herbs (CH) to Manage Cancer-related Symptoms in Patients With Advanced Non-small-cell- Lung Cancer (NSCLC)
Brief Title: A Feasibility Study of Chinese Herbs to Manage Cancer-related Symptoms in Patients With Advanced NSCLC
Acronym: CH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Thomas Jagoe, MD, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JGH-14-150
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
Keywords: Chinese herbs; lung cancer; quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a feasibility study designed to see if the main study can be done.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chinese herbs formula: Shu Yu Wan (Experimental): All participants will be offered the choice of taking the CH formula in capsules or sachets in addition to standard care. This study will use the Shu Yu Wan formula which comprises 23 different herbs and is based on the best evidence in the literature of use of CH in lung cancer.
  Interventions: Dietary Supplement: Chinese herbs formula: Shu Yu Wan

INTERVENTIONS:
Dietary Supplement: Chinese herbs formula: Shu Yu Wan — The patients will be offered the choice of taking the CH formula in capsules or sachets and given instructions about recommendations to improve palatability. The formula should be taken with meals 3 times a day (each dose is either 1 sachet or 4 capsules) for six-weeks.
  Other Names: Chinese Yam Pill

SUMMARY:
The current proposal is a feasibility and acceptability study to establish the necessary groundwork for more detailed investigations into the role of CH in reducing symptoms and improving quality of life in NSCLC patients at the Jewish General Hospital (JGH). A standardized and easily administered form of CH will be used, incorporating a carefully selected combination of herbs designed to alleviate a range of common symptoms suffered by patients with advanced NSCLC.

DETAILED DESCRIPTION:
Patients with advanced NSCLC, in addition to their very poor chances of cure or extended survival, frequently suffer a range of different symptoms related to both their disease and its treatment. As a result there is a pressing need to develop more effective anti-cancer therapies and an imperative to enhance the effects of existing treatments and alleviate symptoms more effectively.

Increasing numbers of patients with cancer are using complementary medicine, including Chinese herbs (CH), and evidence is accumulating from a growing number of laboratory studies and clinical trials, that CH may exert beneficial effects for cancer patients in many ways.

The current proposal is a feasibility and acceptability study to establish the necessary groundwork for more detailed investigations into the role of CH in reducing symptoms and improving quality of life in NSCLC patients at the JGH. A standardized and easily administered form of CH will be used, incorporating a carefully selected combination of herbs designed to alleviate a range of common symptoms suffered by patients with advanced NSCLC.

This is a prospective, longitudinal cohort study of a 6-week clinical intervention with Chinese herbs in advanced (Stage 4) NSCLC patients All the active patients who have histologically or cytologically proven metastatic NSCLC with Eastern Cooperative Oncology Group (ECOG) performance status of 0 -2 will be eligible to participate in the study. Quality of life will be assessed by FACT-L and Edmonton Symptom Assessment System (ESAS) questionnaires. Patient will be instructed to complete a diary each day to confirm adherence to treatment and to indicate the reason(s) that any doses were missed or treatment was stopped.

ELIGIBILITY:
Inclusion Criteria:

* Stages 4
* ECOG performance ≤ 3
* Life expectancy greater than ≥ 3 months

Exclusion Criteria:

* Receiving Tyrosine Kinase Inhibitors (TKI), (Tarceva, Iressa)
* Brain metastases
* Patients or families who do not speak English or French
* Abnormal liver function: Alanine aminotransaminase (ALT) > 40 U/L, Aspartate aminotransaminase (AST) > 55 U/L, Alkaline phosphatase (ALP) > 145 U/L , Bilirubin > 1.7 umol/L.
* Taking regular anti-convulsants, Coumadin or related anti-coagulant, lithium
* Taking regular immunosuppressive medications: azathioprine (Imuran), basiliximab (Simulect), cyclosporine (Neoral, Sandimmune), daclizumab (Zenapax), muromonab-CD3 (OKT3, Orthoclone OKT3), mycophenolate (CellCept), tacrolimus (FK506, Prograf), sirolimus (Rapamune)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jagoe, MD, Principal Investigator — Lady Davis Institute
Locations (1):
- Peter Brojge Lung Cancer Center, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed journal
Supporting Information: CSR
Time Frame: 2019-08-20
Access Criteria: 1. Kasymjanova G, Tran AT, Cohen V, Pepe C, Sakr L, Small D, Agulnik JS, Jagoe RT: The use of a standardized Chinese herbal formula in patients with advanced lung cancer: a feasibility study. Journal of integrative medicine 2018, 16(6):390-395.
URL: https://www.ncbi.nlm.nih.gov/pubmed/30292672

RESULTS

PARTICIPANT FLOW:
Groups:
- Chinese Herbs Formula: A single-arm, prospective study design was chosen to test the feasibility and acceptability of using the selected Chinese herbs (CH) formula in patients with stage 4 non-small cell lung cancer (NSCLC). All participants will be offered the choice of taking the CH formula in capsules or sachets in addition to standard of care. The formula should be taken with meals 3 times a day (each dose is either 1 sachet or 4 capsules) for 6 weeks.
Period: Overall Study
Arm/Group | Chinese Herbs Formula
Started (In the absence of prior data to guide formal power calculations, a sample size of 15 was chosen.) | 15
Completed | 14 (14 patients, 1 dropped out)
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Chinese Herbs Formula: Shu Yu Wan: All participants will be offered the choice of taking the CH formula in capsules or sachets in addition to standard care. This study will use the Shu Yu Wan formula which comprises 23 different herbs and is based on the best evidence in the literature of use of CH in lung cancer. The formula should be taken with meals 3 times a day (each dose is either 1 sachet or 4 capsules) for six-weeks.
Arm/Group | Chinese Herbs Formula: Shu Yu Wan
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the time of enrollment treated as a continues variable
  years | 63 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Number; unit: participants] — Body mass index measured at the baseline and categorized as:
  Low <19.5 kg/m2 Normal 19.6-24.5 kg/m2 High >24.6 kg/m2
  participants
    Low (<19.5) | 2
    Normal (19.6-24.5) | 8
    High (>24.5) | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Grade ECOG 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  participants
    ECOG PS 0-1 | 12
    ECOG PS 2-3 | 3
Smoking status [Number; unit: participants] — Smokers had a history of consuming at least 5 cigarettes a day in the last 2 years; Ex-smokers are those who quit smoking 2 or more years ago; Non-smoker are those who never smoke a cigarette during the life time. Fo purpose of this study participants categorized as ex/never smokers versus smokers
  participants
    Ex/never smoker | 14
    Smoker | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Using CH for Full-scale Future Research
Description: Number of participants consented over the total number of approached for the study.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- A Single Arm, Prospective Study: Participants received CH formula in 1 sachet or 4 capsules 3 times a day for 6 weeks
Arm/Group | A Single Arm, Prospective Study
Number analyzed (Participants) | 26
participants
  enrolled | 15
  refused | 6
  already taking some herbal supplement | 5

2. Secondary Outcome: Change in QOL From Baseline on the 36 Items Functional Assessment of Cancer Therapy - Lung (FACT-L) at the End of the Study (Week 6)
Description: Functional Assessment of Cancer Therapy - Lung (FACT-L) is a 36-item self-assessment questionnaire that measures QOL over the past week in patients with lung cancer. The FACT-L is made up of five subscales of question rated on a five-point Likert scale and include physical well-being (PWB, range of scores is 0-28), social/family well-being (SWB, range of scores is 0-28), emotional well-being (EWB, range of scores is 0-24), functional well-being (FWB, range of scores is 0-28), and symptoms of lung cancer scale (LCS, range of scores is 0-36). For all subscales higher score is better. A total overall score (0-144). Alternative scoring includes the Trial Outcome Index (TOI), which is the sum of the Physical, Functional, and Lung Cancer Subscales. Total score ranges from 0-92 with high score being better. The clinically meaningful changes of this measure is 6 points. Unit measure is scores on a scales.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: The Functional Assessment of Cancer Therapy - Lung (FACT-L) subscales scores. Higher scores is considered better.
- 6 Weeks: Functional Assessment of Cancer Therapy - Lung (FACT-L) subscales scores. Higher score is considered better.
Arm/Group | Baseline | 6 Weeks
Number analyzed (Participants) | 14 | 14
score on a scale
  Physical well-being | 20.6 (5.2) | 23.3 (1.6)
  Social well-being | 20.4 (4.3) | 20.3 (4.7)
  Emotional well-being | 15.8 (5.4) | 16.1 (5.0)
  Functional well-being | 15.9 (5.4) | 17.2 (5.2)
  Lung cancer scale | 17.5 (3.6) | 18.1 (3.8)
  Trial outcome index | 90.2 (17.2) | 93.9 (13.8)
Statistical Analysis 1: Comparison: Baseline; Comparisons of repeated measures were made using paired sample t test, which compared subjects data at 2 different times: baseline and end of the study. A P value of 0.05 was considered statistically significant; Test type: Equivalence — The equivalence assumes that the true mean difference between the paired samples is zero. Under this model, all observable differences are explained by random variation.Equality margins are: Upper Equivalence Margin=1.5 Lower Equivalence Margin=-1.5; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Physical Well-Being Scores at Baseline and 6 Weeks
Description: The Physical well-being (PWB) subscale has 7 questions with the range of the score from 0 to 4 each. The range of the total score is 0 to 28. The higher the score the better the physical well-being. Effect size (ES) of this study based on magnitude difference of PWB scale of the FACT-L between two measures (baseline and 6 weeks). This ES will be used to calculate sample size in Phase 2 study
Time Frame: Baseline and 6 weeks
Population: P value (calculated) =0.03
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; 6 Weeks: Physical Well-Being (PWB) of the Functional Assessment of Cancer Therapy - Lung (FACT-L), range of the score 0-28, with 0 being best and 28 being worse
Arm/Group | Baseline | 6 Weeks
Number analyzed (Participants) | 14 | 14
score on a scale | 20.6 (5.2) | 22.3 (1.6)

4. Secondary Outcome: Safety of Using Chinese Herb Formula in Patients With Advanced NSCLC
Description: Presence of new symptoms or changes in blood tests suggestive of new toxicity based on Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: Baseline and 6 weeks
Population: Number of adverse events reported between baseline and 6 weeks
Measure: Number; unit: reported adverse events
Groups:
- A Single Arm, Prospective Study: A single-arm, prospective study design was chosen to test the feasibility and acceptability of using the selected CH formula in patients with stage 4 NSCLC at our center. Patients with stage 4 NSCLC were eligible if they had Eastern Cooperative Oncology Group performance status of 0-2 and had not used CHs. In addition, to ensure that no CH-related side effects were misattributed to chemotherapy, only patients who had completed at least one cycle of their current standard chemotherapy and were clinically stable were eligible. Patients who were not on treatment were also eligible if there was no plan to recommence the treatment within the next 6 weeks. To safeguard those who were perceived to be potentially at increased risk of side effects from CHs, patients with active brain metastases, abnormal liver function or those taking tyrosine kinase inhibitors, immunosuppressive drugs, anticonvulsant and anticoagulant medications were excluded.
Arm/Group | A Single Arm, Prospective Study
Number analyzed (Participants) | 15
reported adverse events
  Total number of reported adverse events (AE) | 26
  Grade 1 AEs | 22
  Grade 2 AEs | 4
  Related to CH fomula | 3

5. Secondary Outcome: Change From the Baseline in Symptoms on the Edmonton Symptom Assessment System (ESAS)
Description: The Edmonton Symptom Assessment System (ESAS) is a valid and reliable assessment tool to assist in the assessment of common symptoms experienced by cancer patients including: sleep, well-being, pain, strength, appetite, nausea, vomiting, constipation, drowsiness, tiredness, shortness of breath, depression, anxiety, and distress. Each symptom is rated from 0 to 10 cm on a numerical scale; with 0 meaning that the symptom is absent and 10 that it is the worst possible severity.
Time Frame: Baseline and 6 weeks
Population: P value calculated
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; 6 Weeks: Edmonton Symptom Assessment System
Arm/Group | Baseline | 6 Weeks
Number analyzed (Participants) | 14 | 14
score on a scale
  Sleep | 3.0 (3.2) | 2.9 (1.9)
  Well-being | 3.7 (2.1) | 2.3 (1.5)
  Pain | 2.2 (2.2) | 1.7 (2.0)
  Strength | 4.2 (2.5) | 3.4 (2.4)
  Appetite | 3.1 (3.2) | 2.4 (2.1)
  Nausea | 1.7 (2.4) | 0.8 (1.5)
  Vomiting | 0.5 (1.4) | 0.6 (1.3)
  Constipation | 1.5 (2.6) | 1.4 (2.4)
  Drowsiness | 3.2 (2.8) | 1.8 (2.0)
  Tiredness | 4.0 (2.8) | 2.8 (2.7)
  Shortness of breath | 3.1 (3.0) | 2.8 (2.7)
  Depression | 21 (1.9) | 2.3 (2.3)
  Anxiety | 2.8 (2.6) | 2.5 (2.1)
  Distress | 2.4 (2.5) | 2.3 (2.5)
Statistical Analysis 1: Comparison: Baseline vs 6 Weeks; Test type: Superiority — Pared t-test was used to evaluate the significance of the change in scores; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: not different
Arm/Group | A Single Arm, Prospective Study
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Single Arm, Prospective Study (N=15)
Nausea (Gastrointestinal disorders) | 5 (5) — Intermittent
constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Loss of appetite (Gastrointestinal disorders) | 3 (3)
Infections (Infections and infestations) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Dermatitis (Musculoskeletal and connective tissue disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This is a small study in a single centre leading to small number of subjects Caveat: further randomized controlled study needed to confirm the safety and benefit of of CH formula.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02331394/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT02331394/SAP_001.pdf
  • Informed Consent Form (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02331394/ICF_002.pdf